CLINICAL TRIAL: NCT02171975
Title: A Comparison of Conventional Landmark Guided Midline Versus Pre-procedure Ultrasound - Guided Paramedian Techniques in Spinal Anesthesia
Brief Title: Ultrasound - Guided Paramedian Techniques in Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Karthikeyan Kallidaikurichi Srinivasan, Specialist Registrar,Anaesthetics,Cork University Hospital, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECM 4(j) 04/02/14
Record Dates: First submitted 2014-06-19; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Anaesthesia
Keywords: Spinal anaesthesia; Ultrasound pre-procedure guided; Paramedian spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group C (Active Comparator): Patients in this group underwent Conventional landmark guided midline spinal anaesthetic.
  Interventions: Procedure: Conventional landmark guided midline spinal anaesthetic
- Group P (Experimental): This group had their spinal anaesthetic done based on pre-procedure ultrasound guided paramedian spinal
  Interventions: Procedure: pre-procedure ultrasound guided paramedian spinal

INTERVENTIONS:
Procedure: pre-procedure ultrasound guided paramedian spinal — In group P, a portable ultrasound unit was used for initial pre-procedural marking. The interspinous space at which the clearest image of the anterior complex (ligamentum flavum dura complex- LFD) and posterior complex (posterior longitudinal ligament- PLL) was obtained, was selected. At the selected interspace, and with the probe positioned to obtain the clearest ultrasound image, a skin marker was used to mark the midpoint of the long border of the probe and the midpoints of the short borders of the probe . At the same horizontal level as the midpoint of the long border of the probe, the midpoint of the line drawn between the two short border midpoints of the probe was used as paramedian insertion point for the spinal needle.
  Arms: Group P
Procedure: Conventional landmark guided midline spinal anaesthetic — Spinal anaesthesia was administered based on conventional landmark based midline approach.
  Arms: Group C

SUMMARY:
Multiple passes and attempts while administering spinal anesthesia are associated with a greater incidence of post dural-puncture headache, paraesthesia and spinal hematoma. The investigators hypothesised that the routine use of pre-procedural ultrasound-guided paramedian spinals reduces the number of passes required to achieve enter the subarachnoid space when compared to the conventional landmark-guided midline approach.

DETAILED DESCRIPTION:
Spinal anesthesia is widely performed using a surface landmark based 'blind' technique. Multiple passes and attempts while administering spinal anesthesia are associated with a greater incidence of post dural-puncture headache, paraesthesia and spinal hematoma.

Real time and pre-procedural neuraxial ultrasound techniques have been used to improve the success rate of spinal anesthesia. The use of real time ultrasound-guided spinal anesthesia has to date been limited to case series and case reports. Its use may be limited by the requirement for wide bore needles and the technical difficulties associated with simultaneous ultrasound scanning and needle advancement. The use of pre-procedural ultrasound has been shown to increase the first pass success rate for spinal anesthesia only in patients with difficult surface anatomic landmarks.No technique has been shown to improve the success rate of dural puncture when applied routinely to all patients.

Studies on pre-procedural ultrasound-guided spinal techniques are limited to a midline approach using a transverse median view (TM). The parasagittal oblique (PSO) view consistently offers better ultrasound view of the neuraxis compared to TM views. However no studies have been conducted to assess whether these superior PSO views translate into easier paramedian needle insertion.

We hypothesised that the routine use of pre-procedural ultrasound-guided paramedian spinal technique results in less number of passes required to enter the subarachnoid space when compared to the conventional landmark based midline approach.

ELIGIBILITY:
Inclusion Criteria:

* all consented patients scheduled to undergo elective total knee or total hip arthroplasty under spinal anesthesia were included in the study.

Exclusion Criteria:

* Patients with contraindications to spinal anesthesia (allergy to local anesthetic, coagulopathy, local infection and indeterminate neurological disease) were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of passes | Up to 45 minutes from the start of insertion of spinal needled for administration of spinal anaesthetic
  The number of passes, defined as the number of forward advancements of the spinal needle in a given interspinous space (i.e. withdrawal and redirection of spinal needle without exiting the skin)

SECONDARY OUTCOMES:
Number of spinal needle insertion attempts | Up to 45 minutes from the start of insertion of spinal needled for administration of spinal anaesthetic
  number of spinal needle insertion attempts (defined as the number of times the spinal needle was withdrawn from the skin and reinserted) were noted
Blood in spinal needle | Up to 45 minutes from the start of insertion of spinal needled for administration of spinal anaesthetic
  Presence of blood in spinal needle
Time for identifying landmarks | Up to 10 minutes fraom start of plapating for landmarks - Completed once anethetist declares that markings are complete
  Time for identifying landmarks in group C was defined as time from which the anesthesiologist started palpating to identify the landmarks to completion of the process as declared by the anesthesiologist. In group P it was defined as time from which the ultrasound probe was placed on the skin to the anesthesiologist declaring that the markings are completed
Time taken for performing spinal anesthetic | Up to 45 minutes from the start of insertion of spinal needled for administration of spinal anaesthetic
  defined as time taken from insertion of introducer needle to completion of injection
Incidence of radicular pain | Up to 24 hours after administration of spinal anaesthetic
  Shooting pain going down along one of the dermatomal levels in the leg
Presence of paresthesia | Up to 24 hours after administration of spinal anaesthetic
  Paresthesia along dermatomal distribution during performing spinal anaesthetic
Grading of palpated landmarks | Up to 10 minutes fraom start of plapating for landmarks - Completed once anethetist declares that markings are complete
  Anesthesiologist palpated the landmarks after positioning and graded the ease of palpation on a 4 point scale (easy, moderate, difficult or impossible)
Peri-procedural VAS scores of pain at injection site | up to 30 minutes following spinal anaesthetic injection and prior to sedation
  After positioning and prior to administration of sedation, patients were asked for their peri-procedural pain scores measured using an 11 point verbal rating scale (0=no pain, 10=most pain imaginable)
peri-procedural discomfort scores | up to 30 minutes following spinal anaesthetic injection and prior to sedation
  peri-procedural discomfort scores measured using an 11 point verbal rating measured (0= no discomfort, 10=most discomfort imaginable).
Level of block | 15 minutes after spinal anaesthetic injection
  Dermatomal level at which loss of cold sensation (ethyl chloride spray) occurs

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan Kallidaikurichi Srinivasan, FCARCSI,MD, Principal Investigator — Cork University Hospital
Locations (1):
- South Infirmary Victoria University Hospital, Cork, Cork, Ireland